CLINICAL TRIAL: NCT07406438
Title: An Open-label, Multicenter, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of GB10 Intravitreal Injection in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Brief Title: To Evaluate the Safety, Pharmacokinetics, and Efficacy of GB10 Intravitreal Injection in Patients With Neovascular Age-related Macular Degeneration (nAMD)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Kexing Pharmaceutical Co., Ltd. (Network)
Responsible Party: Sponsor
Organization: Kexing Biopharm Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KXZY-GB10-101
Record Dates: First submitted 2026-01-30; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD)
Keywords: nAMD; GB10; PK/PD

STUDY DESIGN:
Intervention Model Description: nAMD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SAD Dose 1 (Experimental): SAD Dose 1 IVT
  Interventions: Drug: GB10
- SAD Dose 2 (Experimental): SAD Dose 2 IVT
  Interventions: Drug: GB10
- SAD Dose 3 (Experimental): SAD Dose 3 IVT
  Interventions: Drug: GB10
- SAD Dose 4 (Experimental): SAD Dose 4 IVT
  Interventions: Drug: GB10
- SAD Dose 5 (Experimental): SAD Dose 5 IVT
  Interventions: Drug: GB10
- SAD Dose 6 (Experimental): SAD Dose 6 IVT
  Interventions: Drug: GB10
- MAD Dose 1 (Experimental): MAD Dose 1 IVT
  Interventions: Drug: GB10
- MAD Dose 2 (Experimental): MAD Dose 2 IVT
  Interventions: Drug: GB10

INTERVENTIONS:
Drug: GB10 — GB10 Intravitreal Injection with indicating dosage.

SUMMARY:
This study aims to preliminarily evaluate the efficacy and safety of GB10 intravitreal (IVT) injection for the treatment of patients with neovascular age-related macular degeneration (nAMD). It consists of two parts, single-ascending-dose escalation (SAD) and multiple-ascending-dose escalation (MAD).

In SAD, a single IVT of up to 6 doses will be administered to up to 36 treatment-naïve or previously treated patients with nAMD. If the lowest dose is considered safe without dose-limiting toxicity, escalation will proceed to the next higher dose level. At the end of SAD, the two doses that best balance efficacy and safety will be selected and entered into MAD.

In MAD, a single IVT of 2 doses will be administered to 12 treatment-naïve or previously treated patients with nAMD, who will be enrolled across the low- to high-dose levels.

After GB10 intervention, the participants will undergo tests to evaluate the PK/PD characteristics of GB10 and ocular and non-ocular safety.

DETAILED DESCRIPTION:
This is an open-label, multicenter, dose-escalating study in patients with nAMD. The study consists of two parts: single-ascending-dose escalation (SAD) and multiple-ascending-dose escalation (MAD). It aims to evaluate the safety, tolerability, and PK/PD profile of single and multiple GB10 IVT injections in patients with nAMD, to investigate the efficacy of GB10, and to assess its immunogenicity.

In SAD, a single IVT of 6 doses (per-eye administration, the same below) will be administered to up to 36 treatment-naïve or previously treated patients with neovascular age-related macular degeneration (nAMD). Participants will be enrolled sequentially, starting with the lowest dose and progressing to the highest. The first participant of each cohort will serve as the sentinel participant. If no dose-limiting toxicities related to GB10 treatment are observed among the participants, escalation will proceed to the next higher dose level after approval from the safety review committee. Two doses, best balancing efficacy and safety, will be determined in SAD and then entered into MAD.

In MAD, a single IVT of 2 doses will be administered to 12 treatment-naïve or previously treated patients with nAMD, who will be enrolled across the low- to high-dose levels.

After GB10 intervention, the participants will undergo tests to evaluate the PK/PD characteristics of GB10 and ocular and non-ocular safety.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosed with choroidal neovascularization (CNV) secondary to AMD (nAMD); For the study eye, either no prior IVT anti-VEGF treatment (treatment-naïve patients) or the last injection of the prior IVT anti-VEGF treatment occurred > 3 months before the first dose, with investigator-assessed effectiveness of prior anti-VEGF therapy (previously treated patients).
2. The study eye must have either subfoveal CNV or juxtafoveal CNV with a subfoveal component related to the CNV activity (as evidenced by subretinal fluid, subretinal hyper-reflective material, leakage, or hemorrhage);
3. CNV lesion of all types (CNV lesion types in the study eye include predominantly classic, minimally classic, or occult [including polypoidal choroidal vasculopathy (PCV)]) with:

   1. Total lesion size (including blood, atrophy, fibrosis, and neovascularization) of ≤ 9 disc areas by FFA;
   2. CNV component area of ≥ 50% of total lesion size by FFA;
   3. Active CNV confirmed by FFA (evidence of leakage);
   4. CNV exudation confirmed by SD-OCT (presence of fluid).
4. BCVA letter score in the study eye of 78-24 letters (inclusive) in ETDRS-like charts (20/32-20/320 Snellen equivalent) before the first dose;
5. Willingness to participate in the study, to comply with the study protocol, and to provide signed informed consent.

Key Exclusion Criteria:

1. CNV in the study eye due to causes other than AMD, such as ocular histoplasmosis, trauma, pathological myopia, angioid streaks, choroidal rupture, or uveitis;
2. The study eye on FFA:

   1. Subretinal hemorrhage of > 50% of the total lesion area and/or that involves the fovea; or
   2. Fibrosis or atrophy of > 50% of the total lesion area and/or that involves the fovea;
3. Any concurrent intraocular condition in the study eye (e.g., central serous chorioretinopathy [CSC], retinal pigment epithelial tear involving the macula, amblyopia, aphakia, retinal detachment, cataract, diabetic retinopathy or maculopathy, epiretinal membrane with traction, retinal vein occlusion, etc.) that, in the opinion of the investigator, may either reduce the potential for visual improvement or require medical or surgical intervention;
4. Spherical equivalent of the refractive error demonstrating more than 8 diopters of myopia in the study eye (for study eye with prior refractive surgery or cataract surgery, preoperative refractive error demonstrating more than 8 diopters), or axial length >26.5 mm when reliable refractive assessment is unavailable;
5. Uncontrolled glaucoma (e.g., progressive loss of visual fields or defined as IOP≥25 mmHg despite treatment with anti-glaucoma medication) in the study eye;
6. Current or prior receipt of any treatment for the study eye, including but not limited to:

   1. IVT implantation or injection other than anti-VEGF drugs within 6 months before screening (e.g., steroids, transplasminogen activator, ocriplasmin, C₃F₈ gas, air filling);
   2. Periocular pharmacological interventions for retinal diseases within 6 months before screening (including subconjunctival, sub-tenon's, peribulbar, or retrobulbar injections);
   3. Laser/photodynamic therapies within 6 months before screening (including laser photocoagulation, verteporfin PDT, diode laser, or transpupillary thermotherapy);
   4. Cataract surgery within 3 months before screening, or corticosteroid treatment for complications of cataract surgery, or YAG (yttrium aluminum garnet) laser posterior capsulotomy;
   5. Prior other intraocular surgery (e.g., pars plana vitrectomy [PPV], glaucoma surgery [except YAG peripheral iridotomy >3 months prior], corneal transplant, or radiotherapy).
7. Active intraocular inflammation (grade trace or above) in the study eye before the first dose;
8. Current vitreous hemorrhage (grade trace or above) in the study eye before the first dose;
9. Monocular vision or non-study eye BCVA < 24 letters before the first dose;
10. History of any cardiovascular/cerebrovascular events within 6 months before the first dose, including but not limited to: stroke (cerebrovascular accident), myocardial infarction, unstable angina, ventricular arrhythmias, and heart failure ≥ NYHA Class II;
11. History of major surgery within 6 months before the first dose or plan to undergo surgery during the study;
12. History of other disease, metabolic dysfunction, abnormal physical examination finding, or clinical laboratory finding prompting reasonable suspicion of a condition that might affect interpretation of the results of the study or render the patient at high risk for treatment complications in the opinion of the investigator, including but not limited to:

    1. Hepatic/renal dysfunction (ALT/AST>2.5×ULN; Cr/BUN>2×ULN);
    2. Uncontrolled diabetes (HbA1c≥7.5%);
    3. Uncontrolled hypertension (resting SBP ≥160 mmHg and/or DBP ≥100 mmHg);
    4. Platelets<100×10⁹/L; or coagulation dysfunction (PT>3 sec above ULN; APTT >10 sec above ULN);
13. Pregnant or nursing (lactating) women;
14. Any other conditions deemed by the investigator to render the participant unsuitable for trial participation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of ocular adverse events | From enrollment to the end of treatment at 12 weeks
The incidence and severity of non-ocular adverse events | From enrollment to the end of treatment at 12 weeks
(SAD) The change in best corrected visual acuity (BCVA) from baseline after 4 weeks of treatment | From enrollment to the end of treatment at 4 weeks
(MAD) The change in best corrected visual acuity (BCVA) from baseline after 12 weeks of treatment | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
(SAD) Change in central retinal subfield thickness (CST) from baseline at 4 weeks of treatment | From enrollment to the end of treatment at 4 weeks
(MAD) Change in central retinal subfield thickness (CST) from baseline at 12 weeks of treatment | From enrollment to the end of treatment at 12 weeks
Time of receiving rescue therapy for nAMD activity | From enrollment to the end of treatment at 12 weeks
Positive rate of anti-drug antibody and neutralizing antibody of GB10 | From enrollment to the end of treatment at 12 weeks
Area under the drug-time curve from 0 to time t of GB10 | From enrollment to the end of treatment at 12 weeks
Area under the curve at the time of 0-infinity of GB10 | From enrollment to the end of treatment at 12 weeks
Peak concentration of GB10 | From enrollment to the end of treatment at 12 weeks
Peak time of GB10 | From enrollment to the end of treatment at 12 weeks
Clearance rate of GB10 | From enrollment to the end of treatment at 12 weeks
Half-life of GB10 | From enrollment to the end of treatment at 12 weeks
VEGF concentration | From enrollment to the end of treatment at 12 weeks
Ang2 concentration | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Henan Provincial Eye Hospital, Zhengzhou, Henan
  - Nanchang University Second Affiliated Hospital, Nanchang, Jiangxi
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital (SRRSH), affiliated with Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No